CLINICAL TRIAL: NCT00020566
Title: European Ewing Tumour Working Initiative of National Groups Ewing Tumour Studies 1999 (EURO-E.W.I.N.G.99)
Brief Title: Combination Chemotherapy With or Without Peripheral Stem Cell Transplantation, Radiation Therapy, and/or Surgery in Treating Patients With Ewing's Sarcoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Cancer and Leukaemia Group (Other); Societe Francaise Oncologie Pediatrique (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network); German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other); Gesellschaft fur Padiatrische Onkologie und Hamatologie - Austria (Other); Swiss Cancer Institute (Other); EBMT Solid Tumors Working Party (Other); Children's Oncology Group (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068608; EURO-EWING-INTERGROUP-EE99; EBMT-INTERGROUP-EE99; EORTC-62981; GPOH-AUSTRIA-INTERGROUP-EE99; GPOH-GERMANY-INTERGROUP-EE99; SFOP-INTERGROUP-EE99; SWS-SAKK-INTERGROUP-EE99; CCLG-INTERGROUP-EE99; COG-AEWS0331; EU-20213
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2012-06

CONDITIONS: Sarcoma
Keywords: localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Dactinomycin; Busulfan; Doxorubicin; Etoposide; Ifosfamide; Melphalan; Vincristine; Radiotherapy

ARMS (3):
- Group 1 (Experimental): Patients receive 2 additional courses of VIDE induction chemotherapy (courses 5 and 6). Patients requiring radiotherapy to the axial tumor also undergo concurrent radiotherapy 5 days a week. Some patients may then undergo surgical resection of the tumor. All patients will then receive vincristine IV on day 1 and dactinomycin IV and ifosfamide IV over 3 hours on days 1 and 2 (VAI). Treatment repeats every 21 days for 8 courses (courses 7-14). Patients requiring radiotherapy to the brain and/or spinal cord also undergo concurrent radiotherapy.
  Interventions: Biological: dactinomycin; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: radiation therapy
- Group 2, arm I (Experimental): Patients undergo 2 additional courses of VIDE induction chemotherapy (courses 5 and 6). Some patients may then undergo surgical resection of the tumor. All patients receive VAI chemotherapy as in group 1 for 1 course. Patients then receive 7 additional courses of VAI chemotherapy (courses 8-14). Patients with unresectable, partially resected, or inadequately resected disease undergo concurrent whole-lung radiotherapy for 6-12 days.
  Interventions: Biological: dactinomycin; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: radiation therapy
- Group 2, arm II (Experimental): Patients undergo 2 additional courses of VIDE induction chemotherapy (courses 5 and 6). Some patients may then undergo surgical resection of the tumor. All patients receive VAI chemotherapy as in group 1 for 1 course. Patients then receive high-dose chemotherapy comprising oral busulfan every 6 hours on days -6 to -3 and melphalan IV over 30 minutes on day -2. Patients receive autologous PBSC IV on day 0. Patients with unresectable, partially resected, or inadequately resected disease undergo concurrent radiotherapy 5 days a week for at least 5 weeks.
  Interventions: Biological: dactinomycin; Drug: busulfan; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: melphalan; Drug: vincristine sulfate; Procedure: autologous hematopoietic stem cell transplantation; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: dactinomycin — Given IV
Drug: busulfan — Given orally and IV
  Arms: Group 2, arm II
Drug: doxorubicin hydrochloride — Given IV
Drug: etoposide — Given IV
Drug: ifosfamide — Given IV
Drug: melphalan — Given orally and IV
  Arms: Group 2, arm II
Drug: vincristine sulfate — Given IV
Procedure: autologous hematopoietic stem cell transplantation — Given IV
  Arms: Group 2, arm II
Procedure: conventional surgery — Given to patients deemed to require it
Radiation: radiation therapy — Given to patients deemed to require it

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy and kill more tumor cells. It is not yet known if combination chemotherapy is more effective with or without radiation therapy and/or surgery in treating Ewing's sarcoma.

PURPOSE: This randomized phase III trial is studying different combination chemotherapy regimens to see how well they work when given with or without peripheral stem cell transplantation, radiation therapy, and/or surgery in treating patients with Ewing's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the event-free and overall survival of patients with tumor of the Ewing's family treated with standard induction chemotherapy comprising vincristine, dactinomycin, ifosfamide and etoposide (VIDE) followed by consolidation chemotherapy comprising vincristine, dactinomycin, and ifosfamide versus high-dose busulfan and melphalan (Bu-Mel) followed by autologous peripheral blood stem cell (PBSC) transplantation with or without radiotherapy and/or surgery.

Secondary

* Determine the prognostic significance of EWS-Flil transcript in these patients.
* Determine the frequency and prognostic value of minimal disease in bone marrow and PBSC, as determined by the presence or absence of EWS-Flil transcript, in these patients.
* Determine the feasibility and toxicity of VIDE induction chemotherapy in these patients.
* Determine the response of these patients to VIDE induction chemotherapy.
* Determine the feasibility and toxicity of VAI consolodation chemotherapy in these patients.
* Determine the feasibility and toxicity of Bu-Mel consolodation chemotherapy in these patients.
* Determine event-free survival and overall survival of patients treated with these regimens by prognostic group analysis.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age and local treatment of the primary tumor (yes vs no).

Patients receive induction chemotherapy comprising vincristine IV on day 1 and ifosfamide IV over 3 hours, doxorubicin IV over 4 hours, and etoposide IV over 1 hour on days 1-3 (VIDE). Treatment repeats every 21 days for 4 courses in the absence of unacceptable toxicity. Peripheral blood stem cells (PBSC) are collected after course 3 and/or 4. Patients are evaluated after course 4. Patients in need of early radiotherapy due to an axial tumor or patients who require radiotherapy to the brain and/or spinal cord (at any time during study) are assigned to group 1. Patients not needing early radiotherapy are assigned to group 2.

* Group 1: Patients receive 2 additional courses of VIDE induction chemotherapy (courses 5 and 6). Patients requiring radiotherapy to the axial tumor also undergo concurrent radiotherapy 5 days a week. Some patients may then undergo surgical resection of the tumor. All patients will then receive vincristine IV on day 1 and dactinomycin IV and ifosfamide IV over 3 hours on days 1 and 2 (VAI). Treatment repeats every 21 days for 8 courses (courses 7-14). Patients requiring radiotherapy to the brain and/or spinal cord also undergo concurrent radiotherapy.
* Group 2: Patients undergo 2 additional courses of VIDE induction chemotherapy (courses 5 and 6). Some patients may then undergo surgical resection of the tumor. All patients receive VAI chemotherapy as in group 1 for 1 course. Patients are randomized to 1 of 2 consolidation therapy arms.

  * Arm I: Patients receive 7 additional courses of VAI chemotherapy (courses 8-14). Patients with unresectable, partially resected, or inadequately resected disease undergo concurrent whole-lung radiotherapy for 6-12 days.
  * Arm II: Patients receive high-dose chemotherapy comprising oral busulfan every 6 hours on days -6 to -3 and melphalan IV over 30 minutes on day -2. Patients receive autologous PBSC IV on day 0. Patients with unresectable, partially resected, or inadequately resected disease undergo concurrent radiotherapy 5 days a week for at least 5 weeks.

Patients are followed every 3 months for 4 years, every 6 months for 1 year, and then periodically thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: Approximately 1,200 patients will be accrued for this study within approximately 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed tumor of the Ewing's family of bone or soft tissue

  * Ewing's sarcoma
  * Peripheral primitive neuroectodermal tumor
* Disease meeting one of the following criteria:

  * Resectable localized disease (tumor volume less than 200 mL)
  * Localized disease previously resected at diagnosis
  * Unresectable disease (at least 200 mL tumor volume) but radiotherapy as local control can be delayed
  * Localized disease with early radiotherapy required
  * Pulmonary and/or pleural metastases only
  * Extrapulmonary/pleural metastases (skeleton, bone marrow, lymph nodes)
* No more than 45 days since definitive biopsy

PATIENT CHARACTERISTICS:

Age:

* Under 50

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Renal function normal
* Glomerular filtration rate at least 60 mL/min

Cardiovascular:

* Normal cardiac function
* Fractional shortening at least 29%
* Ejection fraction at least 40%

Other:

* No medical, psychiatric, or social condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2001-02; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Event-free survival
Overall survival

SECONDARY OUTCOMES:
Feasibility, toxicity, and response at 1 month following induction therapy
Feasibility and toxicity of consolidation regimens at 1 month following consolidation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alan W. Craft, MD, Study Chair — Sir James Spence Institute of Child Health at Royal Victoria Infirmary; Ian J. Lewis, MD, Study Chair — Leeds Cancer Centre at St. James's University Hospital; Odile Oberlin, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Ian R. Judson, MA, MD, FRCP — Institute of Cancer Research, United Kingdom; Heribert F. Juergens, MD, Study Chair — University Hospital Muenster; Helmut Gadner, MD, FRCPG, Study Chair — St. Anna Kinderkrebsforschung; G. Ulrich Exner, MD, Study Chair — Balgrist Universitaetsklinik; Ruth Ladenstein, MD, Study Chair — St. Anna Kinderkrebsforschung; Douglas Hawkins, MD, Study Chair — Seattle Children's Hospital
Locations (103):
- United States (88):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's Hospital Colorado Center for Cancer and Blood Disorders, Aurora, Colorado
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics of Minnesota - St. Paul, Saint Paul, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (9):
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's and Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- Starship Children's Health, Auckland, New Zealand
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Result] Ladenstein R, Potschger U, Le Deley MC, Whelan J, Paulussen M, Oberlin O, van den Berg H, Dirksen U, Hjorth L, Michon J, Lewis I, Craft A, Jurgens H. Primary disseminated multifocal Ewing sarcoma: results of the Euro-EWING 99 trial. J Clin Oncol. 2010 Jul 10;28(20):3284-91. doi: 10.1200/JCO.2009.22.9864. Epub 2010 Jun 14. PMID 20547982
- [Result] Le Deley MC, Delattre O, Schaefer KL, Burchill SA, Koehler G, Hogendoorn PC, Lion T, Poremba C, Marandet J, Ballet S, Pierron G, Brownhill SC, Nesslbock M, Ranft A, Dirksen U, Oberlin O, Lewis IJ, Craft AW, Jurgens H, Kovar H. Impact of EWS-ETS fusion type on disease progression in Ewing's sarcoma/peripheral primitive neuroectodermal tumor: prospective results from the cooperative Euro-E.W.I.N.G. 99 trial. J Clin Oncol. 2010 Apr 20;28(12):1982-8. doi: 10.1200/JCO.2009.23.3585. Epub 2010 Mar 22. PMID 20308673
- [Result] Juergens C, Weston C, Lewis I, Whelan J, Paulussen M, Oberlin O, Michon J, Zoubek A, Juergens H, Craft A. Safety assessment of intensive induction with vincristine, ifosfamide, doxorubicin, and etoposide (VIDE) in the treatment of Ewing tumors in the EURO-E.W.I.N.G. 99 clinical trial. Pediatr Blood Cancer. 2006 Jul;47(1):22-9. doi: 10.1002/pbc.20820. PMID 16572419
- [Derived] Stork T, Ranft A, Aigner C, Jurgens H, Ladenstein RL, Timmermann B, Van den Berg H, Dirksen U, Collaud S. Primary Mediastinal Ewing's Sarcoma: Post Hoc Analysis from Two International Multicenter Prospective Randomized Trials. Cancers (Basel). 2025 Jan 2;17(1):118. doi: 10.3390/cancers17010118. PMID 39796745
- [Derived] Rechl V, Ranft A, Bhadri V, Brichard B, Collaud S, Cyprova S, Eich H, Ek T, Gelderblom H, Hardes J, Haveman LM, Hartmann W, Hauser P, Heesen P, Jurgens H, Kanerva J, Kuhne T, Raciborska A, Rascon J, Streitburger A, Uhlenbruch Y, Timmermann B, Kersting J, Pham MT, Dirksen U. Factors Influencing the Outcome of Patients with Primary Ewing Sarcoma of the Sacrum. Sarcoma. 2024 Mar 16;2024:4751914. doi: 10.1155/2024/4751914. eCollection 2024. PMID 38524902
- [Derived] Corvest V, Marec-Berard P, Lervat C, Pacquement H, Toulmonde M, Gentet JC, Laurence V, Cleirec M, Mansuy L, Bompas E, Castex MP, Taque S, Filhon B, Tabone MD, Verite C, Entz-Werle N, Saumet L, Guimard G, Pondrom M, Chevreau C, Flandrin J, Duranteau L, Rousset-Jablonski C, Brugieres L, Jimenez M, Le Deley MC, Gaspar N, Fresneau B. Late toxicity comparison of alkylating-based maintenance regimen with cyclophosphamide (VAC) vs ifosfamide (VAI) in Ewing sarcoma survivors treated in the randomized clinical trial Euro-EWING99-R1 in France. Int J Cancer. 2023 Apr 15;152(8):1659-1667. doi: 10.1002/ijc.34326. Epub 2022 Oct 31. PMID 36250317
- [Derived] Dirksen U, Brennan B, Le Deley MC, Cozic N, van den Berg H, Bhadri V, Brichard B, Claude L, Craft A, Amler S, Gaspar N, Gelderblom H, Goldsby R, Gorlick R, Grier HE, Guinbretiere JM, Hauser P, Hjorth L, Janeway K, Juergens H, Judson I, Krailo M, Kruseova J, Kuehne T, Ladenstein R, Lervat C, Lessnick SL, Lewis I, Linassier C, Marec-Berard P, Marina N, Morland B, Pacquement H, Paulussen M, Randall RL, Ranft A, Le Teuff G, Wheatley K, Whelan J, Womer R, Oberlin O, Hawkins DS; Euro-E.W.I.N.G. 99 and Ewing 2008 Investigators. High-Dose Chemotherapy Compared With Standard Chemotherapy and Lung Radiation in Ewing Sarcoma With Pulmonary Metastases: Results of the European Ewing Tumour Working Initiative of National Groups, 99 Trial and EWING 2008. J Clin Oncol. 2019 Dec 1;37(34):3192-3202. doi: 10.1200/JCO.19.00915. Epub 2019 Sep 25. PMID 31553693
- [Derived] Le Deley MC, Paulussen M, Lewis I, Brennan B, Ranft A, Whelan J, Le Teuff G, Michon J, Ladenstein R, Marec-Berard P, van den Berg H, Hjorth L, Wheatley K, Judson I, Juergens H, Craft A, Oberlin O, Dirksen U. Cyclophosphamide compared with ifosfamide in consolidation treatment of standard-risk Ewing sarcoma: results of the randomized noninferiority Euro-EWING99-R1 trial. J Clin Oncol. 2014 Aug 10;32(23):2440-8. doi: 10.1200/JCO.2013.54.4833. Epub 2014 Jun 30. PMID 24982464